CLINICAL TRIAL: NCT03843684
Title: Effects of 3D-printed Insoles on Lower Extremity Biomechanics and Knee Joint Loading During Walking and Stair Climbing in Individuals With Knee Osteoarthritis
Brief Title: Effects of 3D-printed on Lower Extremity Biomechanics in Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108DN07
Record Dates: First submitted 2018-12-12; First posted 2019-02-18 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-02

CONDITIONS: Medial Knee Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee osteoarthritis patients (Experimental)
  Interventions: Device: 3D-printed foot orthoses; Device: 5 degrees lateral wedge insoles

INTERVENTIONS:
Device: 3D-printed foot orthoses — 3D printed foot orthoses with arch support
Device: 5 degrees lateral wedge insoles — Insoles with a lateral inclination set at 5 degrees

SUMMARY:
The purposes of this study are: (1) to determine the kinematics, kinetics, and muscle co-activation ratio of level walking and stair negotiation under three different conditions (shoes only, shoes embedded 3D printed insoles, and shoes embedded 5-degree lateral wedges), (2) to build a detailed patient-specific knee model via MR images and musculoskeletal model, then, evaluate the compressive forces acting on the medial aspect of the knee during level walking and stair negotiation.

DETAILED DESCRIPTION:
This study is a cross-sectional study with patients serving as their own control. The investigators will recruit 20 patients with knee osteoarthritis. Using motion capture system, force plates, wireless EMG to capture the motion data of patients during walking and stair negotiation in each condition.

ELIGIBILITY:
Inclusion Criteria:

* Medial knee OA (Kellgren-Lawrence grade I, II or III) according to clinical and radiological criteria of the American College of Rheumatology
* Aged from 50 to 70 years

Exclusion Criteria:

* Neuromuscular illness (e.g., Parkinson disease, Neuropathy)
* Predominant lateral or patella-femoral OA
* Previous of planned hip or knee replacement
* Hip or ankle arthritis
* Rheumatoid arthritis
* Unable to walk without a cane or walker
* Unable to walk up and down the stairs

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Knee adduction moment during level walking and stair negotiation | 10 minutes
  Surrogate marker of medial knee loading. Using motion capture system data to calculate the knee adduction moment via inverse dynamics method.
Medial knee joint contact force during level walking and stair negotiation | 10 minutes
  Calculate the medial knee force to identify the change in medial knee loading by musculoskeletal model. The musculoskeletal model is driven by motion capture system data.
Muscle co-activation ratio during level walking and stair negotiation | 10 minutes
  Level of muscle co-activation measured by electromyography (EMG).

SECONDARY OUTCOMES:
Knee flexion moment during level walking and stair negotiation | 10 minutes
  Surrogate marker of medial and lateral knee loading. Using motion capture system data to calculate the joint moments via inverse dynamics method. The calculated joint moments (N*m) will be normalized by multiplying body weight (Newton) and leg length (meter).
Path of center of pressure during level walking and stair negotiation | 10 minutes
  The factor of affect the joint moments. Measured by force platform.
Lower limbs joint angles during level walking and stair negotiation | 10 minutes
  Lower limbs alignment, including hip, knee and ankle joints. Using motion capture system data to calculate the joint angles.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan